CLINICAL TRIAL: NCT00877851
Title: Development and Evaluation of a Computer-Based, Self-Management Tool for People Recently Diagnosed With Type 2 Diabetes (Evaluation Phase)
Brief Title: Evaluation of a Computer-Based, Self-Management Tool for People With Type 2 Diabetes
Acronym: LWD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Michelle McKinley, Dr Michelle McKinley, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08/NIR01/97
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diet; Physical activity; Self management; Goal setting
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Computer-based Program (Experimental): Use of Computer-based Program for 12 weeks
  Interventions: Behavioral: Computer-based Program
- 2 Control (No Intervention): Usual care and list of useful websites

INTERVENTIONS:
Behavioral: Computer-based Program — The intervention group will receive an initial training session which will include a demonstration of the layout and main features of the computer-based program and some instructions on how to navigate around the different sections of the program. As a minimum level of use, participants will be asked to use the self-monitoring and goal setting aspects of the computer-based program on at least a weekly basis.
  Arms: 1 Computer-based Program

SUMMARY:
NEW Brief Summary: Managing diet and physical activity are vital aspects of diabetes self-care; however, people with diabetes often find it difficult to make changes to their usual diet and physical activity patterns. There is some evidence that computer based education may help some people develop the skills they need to better manage their diabetes. The investigators have developed an external hard drive (a USB stick), focusing on knowledge, self-monitoring, goal setting and skill-development in relation to diet and physical activity for people with Type 2 diabetes. A major emphasis was placed on eliciting the views of people with Type 2 diabetes throughout the development of the computer based program. This study will examine whether this computer based program can improve knowledge, skills and self-care behaviour in people with diabetes. One hundred participants who have been diagnosed with Type 2 diabetes in the past 2 years will be assigned by chance to one of two groups: they will either be assigned to continue with their normal care routine consulting with their doctor as normal, or they will be assigned to use the USB stick at least once a week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of Type 2 diabetes in the past 2 years
* Have access to a computer on a regular basis

Exclusion Criteria:

* Pregnant or lactating
* Other medical conditions where changes in diet or physical activity would be contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle McKinley, PhD, Principal Investigator — Queen's University, Belfast
Locations (2):
- United Kingdom (2):
  - Queen's University Belfast, Belfast, Antrim
  - Belfast Health and Social Care Trust, Belfast, Antrim

REFERENCES:
- [Derived] Booth AO, Lowis C, Hunter SJ, Dean M, Cardwell CR, McKinley MC. Development and Evaluation of a Computer-Based, Self-Management Tool for People Recently Diagnosed with Type 2 Diabetes. J Diabetes Res. 2016;2016:3192673. doi: 10.1155/2016/3192673. Epub 2016 Jun 30. PMID 27446961

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 Computer-based Program | 2 Control
Started | 41 | 43
Completed | 32 | 38
Not Completed | 9 | 5
Not completed — Lost to Follow-up | 5 | 5
Not completed — computer problem | 3 | 0
Not completed — no longer interested in participating | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Computer-based Program | 2 Control | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (9.1) | 60 (10.7) | 59 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 22 | 27 | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Between Group Differences in Diabetes Knowledge
Description: ADKnowl questionnaire
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percent of items correct
Arm/Group | 1 Computer-based Program | 2 Control
Number analyzed (Participants) | 32 | 38
Percent of items correct | 67 (10.4) | 64 (14.2)

2. Primary Outcome: Between Group Differences in Goal Setting
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Between Group Differences in Dietary Intake
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Between Group Differences in Physical Activity Levels
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Between Group Difference in Anthropometry
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Between Group Differences in Markers of Cardiovascular Risk
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Between Group Differences in Markers of Blood Glucose Control
Time Frame: 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Between Group Differences in Self-Efficacy and Barriers to Management of Diabetes
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 1 Computer-based Program | 2 Control
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/43
Other Adverse Events (participants affected / at risk) | 0/41 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes